CLINICAL TRIAL: NCT00002147
Title: Use of Stealth Liposomal Doxorubicin HCl ( DOX-SL ) in the Treatment of Moderate to Severe AIDS-Related Kaposi's Sarcoma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sequus Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 134D; LTI-30-25
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-01

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Liposomes; Doxorubicin; Acquired Immunodeficiency Syndrome; Drug Carriers
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Doxorubicin; Liposomes

INTERVENTIONS:
Drug: Doxorubicin hydrochloride (liposomal)

SUMMARY:
To provide Stealth liposomal doxorubicin hydrochloride ( DOX-SL ) as a therapy for Kaposi's sarcoma patients who have no remaining treatment options other than DOX-SL or patients who have been participating in another DOX-SL protocol and for whom continuation in DOX-SL is medically indicated. Also, to evaluate the safety and efficacy of DOX-SL in patients with Kaposi's sarcoma who have previously received systemic chemotherapy with or without an anthracycline.

DETAILED DESCRIPTION:
Patients receive DOX-SL every 3 weeks for up to 20 cycles.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS-related Kaposi's sarcoma that requires systemic chemotherapy.
* EITHER a medical indication for continuation of DOX-SL following treatment on another DOX-SL protocol, OR no remaining treatment options other than DOX-SL.

Prior Medication:

Allowed:

* Prior anthracyclines.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Cardiac ejection fraction < 50 percent or clinically significant cardiac disease.
* Eligibility for a Liposomal Technology comparative protocol.

Concurrent Medication:

Excluded:

* Other cytotoxic chemotherapy.

Patients with the following prior condition are excluded:

History of idiosyncratic or allergic reaction to anthracyclines.

Prior Medication:

Excluded:

* Chemotherapy within the past 3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Sequus Pharmaceutical Inc, Menlo Park, California, United States

REFERENCES:
- [Background] Jablonowski H, Szelenyi H, Armbrecht C, Mauss S, Niederau C, Strohmeyer G. Liposomal doxorubicin--a new formulation for the treatment of Kaposi's sarcoma: a study on safety and efficacy in AIDS patients. Int Conf AIDS. 1993 Jun 6-11;9(1):397 (abstract no PO-B12-1573)